CLINICAL TRIAL: NCT06723821
Title: Effectiveness of Noninvasive Neuromodulation in Post-COVID Musculoskeletal Pain in the Short Term: Randomized Clinical Trial
Brief Title: Noninvasive Neuromodulation in the Management of Post-COVID Musculoskeletal Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEIM/2022/6/121
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: COVID-19; Musculoskeletal Pain
MeSH Terms: conditions — COVID-19; Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromodulation experimental group (Experimental): The total number of sessions to be carried out on each patient will be 12 sessions, spread over 4 weeks.
  The frequency will be 3 times a week. Each session with NESA microcurrents will last 60 minutes.
  Interventions: Other: Neuromodulation group
- Neuromodulation sham group (Sham Comparator): The total number of sessions to be carried out on each patient will be 12 sessions, spread over 4 weeks.
  The frequency will be 3 times a week. Each session with NESA microcurrents will last 60 minutes.The treatment will be applied with a placebo device that does not emit microcurrent but that has the same function
  Interventions: Other: Neuromodulation sham group

INTERVENTIONS:
Other: Neuromodulation group — During the 12 sessions of which the treatment consists in applying 60 minutes of microcurrent in low intensity.
  Arms: Neuromodulation experimental group
Other: Neuromodulation sham group — During the 12 sessions of which the treatment consists in applying 60 minutes of sham microcurrent in low intensity.
  Arms: Neuromodulation sham group

SUMMARY:
Brief Summary:

The post-Covid syndrome is a problem that affects a significant number of people in the world. Among the most common symptoms is pain, and although there is no specific data on neuropathic pain and Covid, due to under-diagnosis, they may be closely related.

Non-invasive neuromodulation acts on the Central Nervous System through the bioelectrical stimulation of nervous tissue and modulation of the system nervous, and can be useful in acute, chronic and musculosqueletal pain, and in symptoms such as stress, anxiety and sleep disturbances.

The objective of this clinical trial is to assess the efficacy of non-invasive neuromodulation in the treatment of post-Covid musculoskeletal pain. Subjects will be randomly divided into two groups: an experimental group in which non-invasive neuromodulation will be applied and a sham group to which it will be applied off. The variables to be studied before, during and after treatment will be neuropathic pain with the DN4 questionnaire, pain intensity with the EVA scale, sleep quality with the Pittsburgh Sleep Quality Index, level of stress and anxiety with the HADS questionnaire and quality of life with the SF12.

ELIGIBILITY:
Inclusion Criteria:

* Positive result in PCR or antigen test for detecting COVID-19 in the last 3 months.
* Present musculoskeletal pain in the last 3 months.
* Age between 18 to 65 years old.
* Score equal or superior to 4 in DN4 scale.

Exclusion Criteria:

* Present musculoskeletal pain of traumatic origin or known cause
* Present musculoskeletal pain with more than 3 months of evolution.
* Pregnant women
* Present of vascular alterations, malignancy, thrombophlebitis or fever.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Change from Baseline at one month.
  VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health), orientated from the left (worst) to the right (best)

SECONDARY OUTCOMES:
DN4 scale | Change from Baseline at one month.
  It is a clinician-administered questionnaire consisting of 10 items.Seven items related to pain quality (i.e. sensory and pain descriptors) are based on an interview with the patient. These components refer to how the pain feels to the patient Three items are based on the clinical examination. The clinician assesses whether there is reduced sensation (hyposthesia) to touch or pinprick and whether light brushing increases or causes pain (allodynia).The 7 symptoms items are scored by interviewing the patient, and the 3 remaining items are scored by means of clinical examination. The scores are added and a score of 4 or more out of 10 is suggestive of neuropathic pain.
Pittsburg Sleep Quality Index score | Change from Baseline at one month.
  IThe Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality.The scores range from 0 to 21 and the authors suggest that a score >5 be considered as a significant sleep disturbance.
Hospital Anxiety and Depression Scale (HAND) | Change from Baseline at one month
  The HADS is a questionnaire widely used to evaluate anxiety and depression. A 14-item questionnaire to rate patient´s depression and anxiety. Each item has a 0-3 score indicating worse results with higher score
Quality of life SF12 | Change from Baseline at one month.
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure. A higher score is better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pecos-Martin, PhD, Study Director — Alcala University
Locations (1):
- Centro Investigación Fisioterapia y Dolor, Alcalá de Henares, Madrid, Spain